CLINICAL TRIAL: NCT04214002
Title: A Prospective Study to Evaluate the Natural History of Wounds in Patients With Dystrophic Epidermolysis Bullosa (DEB)
Brief Title: The Natural History of Wounds in Patients With Dystrophic Epidermolysis Bullosa (DEB)
Status: Withdrawn | Type: Observational
Why Stopped: Due to the COVID-19 Pandemic, the study was withdrawn.
Sponsor: Krystal Biotech, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: KB-WM-01
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Dystrophic Epidermolysis Bullosa; DEB - Dystrophic Epidermolysis Bullosa
Keywords: DEB; Dystrophic Epidermolysis Bullosa; COL7A1
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a non-interventional, observational study that will evaluate the natural history of wounds in patients with Dystrophic Epidermolysis Bullosa (DEB) for inclusion into the Krystal Biotech Phase III protocol of B-VEC (previously KB103). Wound recurrence and wound size will be evaluated for up to four months.

DETAILED DESCRIPTION:
The objective of this study is to analyze the selected wounds' natural history prior to including the selected wounds in the evaluation of safety and efficacy in Krystal Biotech's Phase III protocol of B-VEC.

Subjects will be enrolled upon obtaining consent and meeting eligibility criteria.

Patient Screening is done on-site, followed by the imaging of at least 1 wound, but up to 15 wounds. All remaining imaging will be performed remotely with a smartphone or tablet application.

Patients are on-trial for approximately four months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is provided. Patients 18 years of age and older, and parent(s)/legal guardian(s) of patients younger than 18 years of age, must provide written informed consent prior to participating in the study; additionally, informed assent will be obtained from patients younger than 18 years of age as specified by local requirements.
* Patient must have a documented diagnosis of DEB based on genetic analysis showing a mutation in COL7A1 or, in the opinion of the investigator, a confirmed diagnosis of DEB based on histologic criteria (antigen mapping or electron microscopy).
* Age: 6 months and older
* Patient must have at least 1 wound that is suitable for imaging, in the opinion of the investigator, at the time of enrollment.
* Patient is willing and able to undergo the protocol-specified procedures.

Exclusion Criteria:

* In the opinion of the investigator, inclusion poses an unacceptable risk to the patient or interpretation of these study data.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients must be 6 months of age or older, and have a diagnosis of DEB based on genetic analysis or histologic criteria. In addition, patients must have at least 1 wound that is suitable for imaging in investigator's opinion at time of screening.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Change in wound surface area | Up to four months
  Percent change in wound surface area from baseline will be measured from images uploaded to an imaging application.

SECONDARY OUTCOMES:
Time to Closure | Up to four months
  The time it takes for a wound to completely close.
Duration of wound closure | Up to four months
  If a closure occurs, the time a wound remains epithelialized after the first, and any subsequent closures.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No